CLINICAL TRIAL: NCT03996525
Title: Electrical Stimulation to Improve Recovery After Peripheral Nerve Injury - A Randomized Controlled Prospective Study
Brief Title: Electrical Stimulation to Improve Recovery After Peripheral Nerve Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Gregory Borschel, MD, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000063546
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hemifacial Paralysis; Bell Palsy
Keywords: unilateral facial nerve palsy; facial nerve palsy; facial palsy; facial paralysis; cross facial nerve graft; CFNG; peripheral nerve stimulation; electrical stimulation; e-stim; free muscle transfer; FMT
MeSH Terms: conditions — Facial Paralysis; Bell Palsy | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation (Experimental): Electrical Stimulation
  The patient will receive active electrical stimulation.
  Interventions: Device: Electrical Stimulation
- Sham Treatment (Placebo Comparator): No Electrical Stimulation
  The patient will receive sham electrical stimulation.
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Electrical Stimulation — Two-Stage Facial Reanimation (Standard Practice) with electrical stimulation for one hour at 20Hz (Experimental Procedure).
  1. Cross-Facial Nerve Graft (CFNG) immediately followed by electrical nerve stimulation proximal to the coaptation site on the donor facial nerve.
  2. Nine-to-Twelve Months later, Free Muscle Transfer (FMT) followed by electrical nerve stimulation proximal to the coaptation site in the intraoral incision.
  Arms: Electrical Stimulation
Device: Sham Treatment — Two-Stage Facial Reanimation (Standard Practice) with sham electrical stimulation for one hour (Placebo).
  1. Cross-Facial Nerve Graft (CFNG) followed by placement of unelectrified electrodes proximal to the coaptation site on the donor facial nerve.
  2. Free Muscle Transfer (FMT) followed by placement of unelectrified electrodes proximal to the coaptation site in the intraoral incision.
  Arms: Sham Treatment

SUMMARY:
After nerve injury and facial palsy, many patients have permanent muscle and sensory dysfunction. Electrical stimulation (ES) of injured nerves may speed up axon growth and improve recovery. This study will assess if ES accelerates motor axon regeneration and improves muscle recovery in patients undergoing two-staged facial reanimation for facial palsy.

This study of ES in these patients will investigate:

i) nerve regeneration over long distances;

ii) direct evidence of changes in nerve regeneration with nerve samples from the second procedure; and

iii) changes in functional outcomes in a patient population with much less variability.

Our study will provide evidence about the effect of ES in improving outcomes in patients with nerve injuries.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing unilateral facial reanimation with a two-stage cross-face nerve graft and free gracilis muscle flap transfer who have;

* i) isolated unilateral facial nerve palsy and
* ii) a functioning contralateral facial nerve.

Exclusion Criteria:

* Any disorders that may compromise nerve regeneration or muscle function following muscle transfer, including diabetes, polyneuropathy, or myopathy and muscular dystrophy.
* Patients with severe cognitive impairment, which would limit their participation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Pre-Operative Lip Excursion with Smile | Change from Baseline (Pre-Op) over 2 Years
  FACEGRAM will be used to objectively analyse change in commissure excursion.
Change in Myelinated Axon Count | Change from Baseline (Pre-Op) to the Final Surgery 1 Year Later
  The number of myelinated nerve fibres that regenerate and reach the distal CFNG will be compared between groups.

SECONDARY OUTCOMES:
Change in Facial Symmetry | Change from Baseline (Pre-Op) over 2 Years
  FACEGRAM will be used to objectively analyse smile symmetry.
Facial Clinimetric Evaluation (FaCE) Scores | Change from Baseline (Pre-Op) Over 2 Years
  The Facial Clinimetric Evaluation (FaCE) Scale is a patient-report questionnaire assessing facial impairment and disability associated with facial paralysis. The 15-item likert scale questionnaire consists of six domains: i) facial movement, ii) facial comfort, iii) oral function, iv) eye comfort, v) lacrimal control and vi) social function.
  Each domain produces its own score, with 1 meaning 'problems all the time' and 5 suggesting 'no problems at all.' The domain scores can then be summed to produce a total score assessing total quality of life with respect to facial paralysis.
Time to Reinnervation | Up to 1 year after the Second Operation (FMT)
  Study participants are requested to monitor their facial movements and record any changes in a daily diary once they first notice facial movement.
Myelin Thickness | Change from Baseline (Pre-Op) to the Final Surgery 1 Year Later
  Using histomorphometry, Myelin Thickness will be used as a surrogate measure for the rate of axon regeneration.
Nerve Fibre Diameter | Change from Baseline (Pre-Op) to the Final Surgery 1 Year Later
  Using histomorphometry, Nerve Fibre Diameter will be used as a surrogate measure for the rate of axon regeneration.
Myelin Thickness/Fibre Diameter Ratio | Change from Baseline (Pre-Op) to the Final Surgery 1 Year Later
  Using histomorphometry, Myelin Thickness/Fibre Diameter Ratio will be used as a surrogate measure for the rate of axon regeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Davidge, MD, Principal Investigator — The Hospital for Sick Children; Ronald Zuker, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada